CLINICAL TRIAL: NCT04113694
Title: Evaluation of Extended Wear Infusion Set (EWIS) in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP298
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Extended Wear Infusion Set (Experimental): Each subject is given 12 Extended Wear Infusion Sets to wear.
  Interventions: Device: Extended Infusion Set

INTERVENTIONS:
Device: Extended Infusion Set — Each subject is asked to wear each Extended Wear Infusion Set for at least 174 hours.
  Other Names: Extended Wear Infusion Set

SUMMARY:
The purpose of this study is to collect confirmatory clinical data to support 6 or 7 days wear of EWIS (Extended Wear Infusion Set).

DETAILED DESCRIPTION:
This study is a multi-center, non-randomized, prospective single arm study with Type 1 patients with diabetes on insulin pump therapy with Continuous Glucose Monitoring (CGM). A total of up to 300 subjects age 18-80 will be enrolled at up to 20 investigational centers in the US. Each subject will wear their own MiniMed™ 670G insulin system. Each subject will be given 12 infusion sets to wear (each infusion set for at least 174 hours, or until infusion set failure if this occurs before 174 hours). Subjects will change insulin reservoirs at least every 174 hours. The time of infusion set insertion will be taken from Daily Log. Subjects can expect to participate for approximately 12-16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 18 - 80 years at the time of screening
2. Subject has type 1 diabetes for more than one year Study specific inclusion criteria
3. Subject is on the MiniMed™ 670G insulin pump therapy within 1 year prior to screening and willing to utilize Auto Mode and CGM with Guardian™ Sensor (3) during the study.
4. Subject is willing and able to perform study procedures as per investigator discretion
5. Subject is willing to take one of the following insulins and can financially support the use of either of the 2 insulin preparations throughout the course of the study (i.e. co-payments for insulin with insurance or able to pay full amount):

   1. Humalog™* (insulin lispro injection)
   2. NovoLog™* (insulin aspart)

Exclusion Criteria:

1. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks.
2. Subject is female and has a positive pregnancy screening test
3. Subject is female of child bearing age and who is sexually active should be excluded if she is not using a form of contraception deemed reliable by investigator
4. Subject is female and plans to become pregnant during the course of the study
5. Subject has Glycosylated hemoglobin (HbA1c) > 8.5 % at time of screening. Note: All HbA1c blood specimens will be sent to and tested by a NGSP certified Central Laboratory. HbA1c testing must follow National Glycohemoglobin Standardization Program (NGSP) standards.
6. Subject has had a history of 1 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to screening

   1. Medical assistance (i.e. Paramedics, Emergency Room [ER] or Hospitalization)
   2. Coma
   3. Seizures
7. Subject has taken any oral, injectable, or IV glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study.
8. Subject is unable to tolerate tape adhesive in the area of infusion set
9. Subject has any unresolved adverse skin condition in the area of infusion set placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection)
10. Subject has infection in the area of infusion set placement at time of screening
11. Subject has had Diabetic Ketoacidosis (DKA) in the 12 months prior to screening visit.
12. Subject is currently abusing illicit drugs
13. Subject is currently abusing alcohol
14. Subject is on dialysis (for renal failure)
15. Subject has history of adrenal disorder
16. Subject has a history of inpatient psychiatric treatment in the past 6 months prior to screening
17. Subject has any condition that the Investigator believes would interfere with study participation
18. Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator
19. Subject has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
20. Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation
21. Subject is using pramlintide (Symlin), SGLT2 inhibitors, GLP agonists, biguanides, DPP-4 inhibitors or sulfonylureas more than 2 weeks from time of screening
22. Subject has been diagnosed with chronic kidney disease requiring dialysis or resulting in chronic anemia
23. Subject has history of cardiovascular disease defined as any ischemic related event or clinically significant arrythmia.
24. Subject has hypothyroidism and has out of reference range thyroid-stimulating hormone (TSH) on screening visit (prior labs in the last 3 months are sufficient). Subject may repeat TSH draw to verify eligibility if not in range

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Medical Investigations, Little Rock, Arkansas
  - AMCR Institute, Escondido, California
  - Stanford University, Palo Alto, California
  - SoCal Diabetes, West Covina, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Metabolic Research Institute, West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Iowa Diabetes and Endocrinology Center, West Des Moines, Iowa
  - Grunberger Diabetes Institute, Bloomfield Hills, Michigan
  - Mayo Clinic (Rochester MN), Rochester, Minnesota
  - Diabetes and Endocrinology Consultants of Pennsylvania, Feasterville-Trevose, Pennsylvania
  - AM Diabetes and Endocrinology Center, Memphis, Tennessee
  - University of Virginia Health System, Charlottesville, Virginia
  - Rainier Clinical Research Center, Renton, Washington

REFERENCES:
- [Derived] Brazg R, Garg SK, Bhargava A, Thrasher JR, Latif K, Bode BW, Bailey TS, Horowitz BS, Cavale A, Kudva YC, Kaiserman KB, Grunberger G, Reed JC, Chattaraj S, Zhang G, Shin J, Chen V, Lee SW, Cordero TL, Rhinehart AS, Vigersky RA, Buckingham BA. Evaluation of Extended Infusion Set Performance in Adults with Type 1 Diabetes: Infusion Set Survival Rate and Glycemic Outcomes from a Pivotal Trial. Diabetes Technol Ther. 2022 Aug;24(8):535-543. doi: 10.1089/dia.2021.0540. Epub 2022 Mar 24. PMID 35263188

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 291 subjects consented and enrolled in the overall study. Of the 291, 28 subjects failed screening, 4 subjects passed screening but did not attempt any EWIS, 259 subjects wore at least one EWIS, 11 subjects early withdraw, 248 subjects completed the study.
Groups:
- Extended Wear Infusion Set: Each subject was given 12 Extended Wear Infusion Sets to wear.
  Extended Infusion Set: each subject was asked to wear each Extended Wear Infusion Set for at least 174 hours.
Period: Overall Study
Arm/Group | Extended Wear Infusion Set
Started | 259
Completed | 248
Not Completed | 11
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 6
Not completed — Withdrawal due to not meeting inclusion and exclusion criteria | 1

BASELINE CHARACTERISTICS:
Groups:
- Humalog Subjects Extended Wear Infusion Set: Each Humalog subject was given 12 Extended Wear Infusion Sets to wear.
  Extended Infusion Set: Humalog subjects were asked to wear each Extended Wear Infusion Set for at least 174 hours.
- Novolog Subjects Extended Wear Infusion Set: Each Novolog subject was given 12 Extended Wear Infusion Sets to wear.
  Extended Infusion Set: Novolog subjects were asked to wear each Extended Wear Infusion Set for at least 174 hours.
- Total: Total of all reporting groups
Arm/Group | Humalog Subjects Extended Wear Infusion Set | Novolog Subjects Extended Wear Infusion Set | Total
Number analyzed (Participants) | 132 | 127 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (14.3) | 46.7 (13.7) | 45.0 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 66 | 134
  Male | 64 | 61 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 126 | 123 | 249
  Unknown or Not Reported | 1 | 0 | 1
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (5.6) | 29.0 (5.9) | 29.0 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Humalog Subjects - Rate of Infusion Set Failure at the End of Day 6
Description: Evaluate rate of infusion set failure due to unexplained hyperglycemia (i.e. suspected occlusion) at the end of Day 6.
Time Frame: 144 hours
Measure: Mean (95% Confidence Interval); unit: Percentage of Extended Wear Infusion Set
Units Other Than Participants: EWIS infusion sets
Groups:
- Extended Wear Infusion Set: Each Humalog subject was given 12 Extended Wear Infusion Sets to wear.
  Extended Infusion Set: Humalog subjects were asked to wear Extended Wear Infusion Set for at least 174 hours.
Arm/Group | Extended Wear Infusion Set
Number analyzed (Participants) | 132
Number analyzed (EWIS infusion sets) | 1561
Percentage of Extended Wear Infusion Set | 0.06 [0.01 to 0.45]

2. Primary Outcome: Novolog Subjects - Rate of Infusion Set Failure at the End of Day 6
Description: Independently evaluate rate of infusion set failure due to unexplained hyperglycemia (i.e. suspected occlusion) at the end of Day 6.
Time Frame: 144 hours
Measure: Mean (95% Confidence Interval); unit: Percentage of Extended Wear Infusion Set
Units Other Than Participants: EWIS infusion sets
Groups:
- Extended Wear Infusion Set: Each Novolog subject was given 12 Extended Wear Infusion Sets to wear.
  Extended Infusion Set: Novolog Subjects were asked to wear each Extended Wear Infusion Set for at least 174 hours.
Arm/Group | Extended Wear Infusion Set
Number analyzed (Participants) | 127
Number analyzed (EWIS infusion sets) | 1480
Percentage of Extended Wear Infusion Set | 0.27 [0.10 to 0.71]

3. Secondary Outcome: Humalog Subject - Rate of Infusion Set Failure at the End of Day 7.
Description: Evaluate rate of infusion set failure due to unexplained hyperglycemia (i.e. suspected occlusion) at the end of Day 7.
Time Frame: 168 hours
Measure: Mean (95% Confidence Interval); unit: Percentage of Extended Wear Infusion Set
Units Other Than Participants: EWIS infusion sets
Groups:
- Extended Wear Infusion Set: Each Humalog subject was given 12 Extended Wear Infusion Sets to wear.
  Extended Infusion Set: Humalog Subjects were asked to wear each Extended Wear Infusion Set for at least 174 hours.
Arm/Group | Extended Wear Infusion Set
Number analyzed (Participants) | 132
Number analyzed (EWIS infusion sets) | 1561
Percentage of Extended Wear Infusion Set | 0.13 [0.03 to 0.51]

4. Secondary Outcome: Novolog Subjects - Rate of Infusion Set Failure at the End of Day 7.
Description: Independently evaluated rate of infusion set failure due to unexplained hyperglycemia (i.e. suspected occlusion) at the end of Day 7.
Time Frame: 168 hours
Measure: Mean (95% Confidence Interval); unit: Percentage of Extended Wear Infusion Set
Units Other Than Participants: EWIS infusion sets
Arm/Group | Extended Wear Infusion Set
Number analyzed (Participants) | 127
Number analyzed (EWIS infusion sets) | 1480
Percentage of Extended Wear Infusion Set | 0.41 [0.16 to 1.00]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Humalog Subjects Extended Wear Infusion Set | Novolog Subjects Extended Wear Infusion Set
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/127
Serious Adverse Events (participants affected / at risk) | 2/132 | 1/127
Other Adverse Events (participants affected / at risk) | 59/132 | 60/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humalog Subjects Extended Wear Infusion Set (N=132) | Novolog Subjects Extended Wear Infusion Set (N=127)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humalog Subjects Extended Wear Infusion Set (N=132) | Novolog Subjects Extended Wear Infusion Set (N=127)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Complication of device removal (General disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 23 (49) | 28 (43)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Infusion site bruising (General disorders) | 0 (0) | 2 (2)
Infusion site cellulitis (Infections and infestations) | 4 (5) | 6 (6)
Infusion site dermatitis (General disorders) | 2 (2) | 1 (1)
Infusion site discomfort (General disorders) | 8 (13) | 6 (6)
Infusion site erythema (General disorders) | 2 (2) | 3 (3)
Infusion site haemorrhage (General disorders) | 0 (0) | 1 (1)
Infusion site hypersensitivity (General disorders) | 1 (3) | 0 (0)
Infusion site infection (Infections and infestations) | 1 (1) | 2 (2)
Infusion site irritation (General disorders) | 0 (0) | 2 (5)
Infusion site nodule (General disorders) | 1 (2) | 2 (2)
Infusion site pain (General disorders) | 4 (7) | 4 (5)
Infusion site reaction (General disorders) | 1 (1) | 0 (0)
Infusion site swelling (General disorders) | 3 (11) | 1 (1)
Infusion site vesicles (General disorders) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medical device site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Medical device site discomfort (General disorders) | 2 (2) | 1 (1)
Medical device site erythema (General disorders) | 1 (1) | 1 (1)
Medical device site irritation (General disorders) | 0 (0) | 1 (1)
Medical device site nodule (General disorders) | 1 (1) | 0 (0)
Medical device site oedema (General disorders) | 0 (0) | 1 (1)
Medical device site swelling (General disorders) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (11) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 2 (3) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tourette's disorder (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT04113694/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT04113694/SAP_001.pdf